CLINICAL TRIAL: NCT01857505
Title: Introduction of the Direct Anterior Approach to Hip Replacement Into a High Volume Community Hospital: Effect on Length of Stay and Hospital Cost
Brief Title: Hip Replacement in a High Volume Community Hospital: Effect on Length of Stay and Hospital Cost
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Anne Arundel Health System Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: IIS-000158
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Hip Osteoarthritis
Keywords: Total Hip replacement; Fracture table; DePuySynthes; Direct anterior approach hip replacement; Posterior approach hip replacement
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Direct Anterior Approach hip replacement: Single surgeon series of 105 consecutive patients who underwent hip replacement via the direct anterior approach on a fracture table
- Posterior Approach Hip Replacement: 105 consecutive patients previously operated on by a less invasive posterior approach at the same institution. These surgeries occurred prior to March, 2010.

SUMMARY:
The investigators propose to evaluate and compare the percentage of patients who are able to be discharged in less than 3 days after undergoing total hip arthroscopy through either a direct anterior or posterior approach, utilizing the identical post operative protocol. The investigators also propose to evaluate the costs associated with the two different approaches to hip replacement in the same group of patients. Post operative resource utilization, discharge disposition, and pain medicine requirement will also be evaluated.

DETAILED DESCRIPTION:
The investigators hypothesize that a higher proportion of patients treated with the direct anterior approach for hip replacement will be able to leave the hospital in less than 3 days when compared with a less invasive posterior approach. Secondly, decreased length of stay associated with the procedure may reduce hospital costs.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive single surgeon series of patients who have undergone primary uncemented hip replacement at our institution through either a posterior approach or direct anterior approach on a fracture table. Posterior approach patient - most recent patient prior to March, 2010, compared with consecutive recent anterior approach patients with minimum of 6 month follow-up.
2. Diagnosis of osteoarthritis, inflammatory arthritis, or avascular necrosis.
3. No previous surgery on affected hip.
4. Age 40-90 at time of surgery

Exclusion Criteria:

1. Patient not permitted to bear full weight after the procedure, per post operative instructions
2. Hip replacement performed for acute fracture.
3. Previous hip surgery.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone primary uncemented hip replacement at our institution (Anne Arundel Medical Center) through either a posterior approach or direct anterior approach on a fracture table utilizing the identical post operative protocol.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | Retrospective review of hospital discharge records
  The length of stay and proportion of patients who went home in less than 3 days will be determined for each group. To evaluate and compare the percentage of patients who are able to be discharged in less than 3 days after undergoing total hip arthroscopy through either a direct anterior or posterior approach, utilizing the identical post operative protocol.
Hospital cost | Retrospective review of utilization records
  Hospital cost analysis will be undertaken for each group.

SECONDARY OUTCOMES:
Post Operative Pain Medication Utilization | After retrospective chart review is complete -- approximately 6 months
  Analysis of post operative pain medicine requirement will be compared for the two groups.
Utilization of inpatient physical therapy resources | Retrospective review -- of hospital discharge
  Utilization of inpatient physical therapy resources and post hospital discharge disposition will be compared for the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul King, M.D., Principal Investigator — Anne Arundel Medical Center / Anne Arundel Orthopedic Surgeons
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

REFERENCES:
- [Background] Hayes JH, Cleary R, Gillespie WJ, Pinder IM, Sher JL. Are clinical and patient assessed outcomes affected by reducing length of hospital stay for total hip arthroplasty? J Arthroplasty. 2000 Jun;15(4):448-52. doi: 10.1054/arth.2000.4346. PMID 10884204
- [Background] Vorhies JS, Wang Y, Herndon J, Maloney WJ, Huddleston JI. Readmission and length of stay after total hip arthroplasty in a national Medicare sample. J Arthroplasty. 2011 Sep;26(6 Suppl):119-23. doi: 10.1016/j.arth.2011.04.036. Epub 2011 Jul 1. PMID 21723700
- [Background] Duwelius PJ, Moller HS, Burkhart RL, Waller F, Wu Y, Grunkemeier GL. The economic impact of minimally invasive total hip arthroplasty. J Arthroplasty. 2011 Sep;26(6):883-5. doi: 10.1016/j.arth.2010.09.011. Epub 2010 Nov 3. PMID 21051190
- [Background] Matta JM, Ferguson TA. The anterior approach for hip replacement. Orthopedics. 2005 Sep;28(9):927-8. doi: 10.3928/0147-7447-20050901-11. No abstract available. PMID 16190055
- [Background] Matta JM, Shahrdar C, Ferguson T. Single-incision anterior approach for total hip arthroplasty on an orthopaedic table. Clin Orthop Relat Res. 2005 Dec;441:115-24. doi: 10.1097/01.blo.0000194309.70518.cb. PMID 16330993